CLINICAL TRIAL: NCT03133923
Title: Safety and Efficacy of Attenuated Mumps Vaccine (Human Diploid Cell)
Brief Title: Phase II of Live Attenuated Mumps (F-genotype) Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Hubei Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015L00195
Record Dates: First submitted 2017-04-17; First posted 2017-04-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Epidemic Parotitis,Mumps
Keywords: Attenuated Mumps Vaccine(F-genotype，Human Diploid Cell, KMB-17), safety, immunogenecity
MeSH Terms: conditions — Mumps | interventions — Mumps Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attenuated Mumps vaccine (KMB-17), low (Experimental): Biological/Vaccine: ≥3.0logCCID50/ml but <3.5 logCCID50/ml Attenuated Mumps vaccine (KMB-17)[ ≥3.0logCCID50/ml but <3.5 logCCID50/ml] in 360 infants (8-24 months old) on 0 day
  Interventions: Biological: ≥3.0 lgCCID50/mlbut <3.5lgCCID50/ml Live Attenuated Mumps Vaccine (Human Diploid Cell) in infants(8-24 months old)
- Attenuated Mumps vaccine (KMB-17), high (Experimental): Biological/Vaccine: ≥4.5logCCID50/ml Attenuated Mumps vaccine (KMB-17)[≥4.5 logCCID50/ml] in 360 infants (8-24 months old) on 0 day
  Interventions: Biological: ≥4.5 lgCCID50/ml Live Attenuated Mumps Vaccine (Human Diploid Cell) in infants(8-24 months old)
- Measles and Mumps Combined Vaccine，Live (Active Comparator): manufacturer：Shanghai Institute of Biological Products Co., Ltd. (SIBP ) Measles and Mumps Combined Vaccine，Live in 360 infants in 360 infants (8-24 months old) on 0 day
  Interventions: Biological: Measles and Mumps Combined Vaccine，Live(SIBP)( positive control)

INTERVENTIONS:
Biological: ≥3.0 lgCCID50/mlbut <3.5lgCCID50/ml Live Attenuated Mumps Vaccine (Human Diploid Cell) in infants(8-24 months old) — ≥3.0 lgCCID50/ml but <3.5lgCCID50/ml;Live Attenuated Mumps (F-genotype) Vaccine (Human Diploid Cell, KMB-17) in 360 infants(aged 8-24 months ) on 0 day
  Arms: Attenuated Mumps vaccine (KMB-17), low
Biological: ≥4.5 lgCCID50/ml Live Attenuated Mumps Vaccine (Human Diploid Cell) in infants(8-24 months old) — ≥4.5CCID50/ml;Live Attenuated Mumps (F-genotype) Vaccine (Human Diploid Cell, KMB-17) in 360 infants(aged 8-24 months ) on 0 day
  Arms: Attenuated Mumps vaccine (KMB-17), high
Biological: Measles and Mumps Combined Vaccine，Live(SIBP)( positive control) — Measles and Mumps Combined Vaccine，Live(SIBP) in 360 infants(aged 8-24 months ) on 0 day
  Arms: Measles and Mumps Combined Vaccine，Live

SUMMARY:
Mumps is an acute infectious respiratory disease caused by the mumps virus (MuV), which occurs mainly in children and adolescents. Its main clinical symptoms were parotid gland suppurative swelling and pain with fever. The pathological changes and harm caused by mumps was not only confined to the parotid gland, on the contrary, the social harm caused by serious complications cannot be ignored. As mumps is a vaccine-preventable infectious disease, vaccination is a fundamental strategy for controlling mumps. So far, there are 13 genotypes of MuV. Based on the analysis of molecular epidemiology, the main epidemic strain of MuV in China was the F genotype. The commonly used vaccine strains represented only a small number of known genotypes, e.g. Jeryl-Lynn (JL) and Rubini strains, which belong to type A, Urabe strain belongs to type B, and L-Zagreb strains belongs to type D. Virus seed of Live Attenuated Mumps Vaccine (Human diploid cell) developed by the institute was SP-A strain, which was the first separation and preparation of the attenuated mumps viruses in China. SP-A belongs to F genotype, which was the domestic epidemic genotype. In addition, the cell substrate prepared for vaccine was human diploid cell (KMB-17 strain), which is much safer to use. The preliminary test results showed that the vaccine possessed good immunogenicity and good antigenic cross-reactivity. The application of this vaccine will provide more effective means to prevent and control of mumps epidemic.

DETAILED DESCRIPTION:
In order to evaluation the safety and immunogenicity of different doses Live Attenuated Mumps Vaccine (Human diploid cell).The study will Determine the optimal dose of vaccine and provide the clinical trail basis for the phase Ⅲ trail design.

Primary objective:

After single dose immunization of low dose(≥3.0but<3.5lgCCID50)、high dose （≥4.5lgCCID50）Live Attenuated Mumps Vaccine (Human Diploid Cell) in Chinese healthy Infants volunteer aged from 8 to 24 months old.the study will evaluate the standardized positive rate of neutralizing antibody and the GMT of the hemagglutination inhibition antibody and neutralizing antibody,proposing the immune reference dose for phase III clinical trials.

Secondary objective： Evaluate the safety of low dose(≥3.0but<3.5lgCCID50)、high dose （≥4.5lgCCID50）Live Attenuated Mumps Vaccine (Human Diploid Cell) in Chinese healthy Infants volunteer aged from 8 to 24 months old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females (from 8 months to 24 months old) as determined by medical history, physical examination, laboratory examination and clinical judgment of the investigator.
* Provided legal identification for the sake of recruitment.
* Without the routine corticosteroids of vaccination .
* Never has gone down with mumps or taken a vaccine contain mumps.
* parent(s)/legal guardian(s) are able to understand and sign informed consents and be able to read a thermometer and dividing ruler .At the same time,the parent(s)/legal guardian(s)should have the ability and objective to comply with the requirements of the protocol.
* Participants or guardians are able to attend all planned clinical appointment and obey and follow all study instructions; can persist for a 1-month visit and receive blood sample and throat swab collection according to program requirements.
* Axillary temperature ≤37℃.

Exclusion Criteria:

* Subject who has a medical history of Mumps or taken a vaccine contain mumps.
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Convulsant,encephalopathy,psychosis or family histoty of epileptics.
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder,it will couse the contraindication of subcutaneous injection
* Any prior administration of attenuated live vaccine in last 15 days;Any prior administration of subunit or inactivated vaccines in last 7 days
* Any prior administration of other research medicines in last 30 days.
* Any prior administration of blood products(immunoglobulin etc.) in last 1 month;Any prior administration of immunodepressant ，cytotoxic drugs or corticosteroids in last 6 months(except the corticosteroids spray can treat irritability rhinitis orcorticosteroids to cure noncomplication acute dermatitis ).
* Any confirmed or suspected autoimmune disease or immune deficiency diseases(like favism or other diseases etc. ), including human immunodeficiency virus (HIV) infection.
* Suffering from congenital deformity or serious chronic disease(congenital heart disease，Down's syndrome,diabetes,sickle cell anemia,nervous illness,cardiocardiopathy,hypertension,bronchitis,pneumonia,asthma,infectious skin diseases)
* Acute or chronic infectious disease,active infectious;Laboratory test show Routine blood abnormal or hepatorenal dysfunction.
* Malignant disease(like cancer)，heredopathia or other disease that will cuase eccyliosis.The spleen or other important organ has been removed for any reason.
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives.

Ages: 8 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1080 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Positive conversion rate of Muv hemagglutination inhibition antibody of different single dose of Muv Vaccine | the 0 days（before vaccination） and 28 day after the vaccination
  To compared the positive conversion rate of Muv hemagglutination inhibition antibody after vaccinate 3 diffirent group (low dose:≥3.0logCCID50/ml but <3.5logCCID50/ml,high dose：≥4.5logCCID50/ml,active comparator :shanghai institute of Biological Products Co,Ltd's measles and Mumps Combined Vaccine.live)
Positive conversion rate of Muv neutralization antibody of different single dose of Muv Vaccine | the 0 days（before vaccination） and 28 day after the vaccination
  To compared the positive conversion rate of Muv neutralization antibody after vaccinate 3 diffirent group (low dose:≥3.0logCCID50/ml but <3.5logCCID50/ml,high dose：≥4.5logCCID50/ml,active comparator :shanghai institute of Biological Products Co,Ltd's measles and Mumps Combined Vaccine.live)

SECONDARY OUTCOMES:
The GMT of the hemagglutination inhibition antibody and neutralizing antibody | the 0 days（before vaccination） and the 28 day after the vaccination
  evaluate the GMT of the hemagglutination inhibition antibody and neutralizing antibody in serum after the subjects get injected different dose of vaccine
The GMT of the neutralizing antibody | the 0 days（before vaccination） and the 28 day after the vaccination
  evaluate the GMT of the neutralizing antibody in serum after the subjects get injected different dose of vaccine
The incidence rate of ADR after vaccination | within the first 28 days after the vaccination
  Study the incidence rate of ADR after vaccination
viral shedding after the vaccination | the 0（before vaccination）,4,10 days after the vaccination
  Using the method of PCR to detection the viral shedding of Muv after the vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Beifang Yang, PhD, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided